CLINICAL TRIAL: NCT01545050
Title: A Phase IIb, Double-Blind, Randomized, Placebo-Controlled, Double-Dummy, Dose-Ranging Study to Evaluate the Clinical Efficacy and Safety of Induction and Maintenance Therapy With BMS-945429 in Subjects With Moderate to Severe Crohn's Disease
Brief Title: Dose Ranging Study of BMS-945429 in Subjects With Moderate to Severe Crohn's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to sponsor decision
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM133-005; 2011-004763-72 (EudraCT Number)
Record Dates: First submitted 2012-03-01; First posted 2012-03-06 (Estimated); Results first posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — clazakizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Induction Cohort: Placebo matching with BMS-945429 (Clazakizumab) (Experimental)
  Interventions: Biological: Placebo matching with BMS-945429
- Induction Cohort: BMS-945429 (Clazakizumab)(600 IV/200 SC mg) (Experimental)
  Interventions: Biological: Placebo matching with BMS-945429; Biological: BMS-945429
- Induction Cohort: BMS-945429 (Clazakizumab)(300 IV/100 SC mg) (Experimental)
  Interventions: Biological: Placebo matching with BMS-945429; Biological: BMS-945429
- Induction Cohort: BMS-945429 (Clazakizumab)(150 IV/100 SC mg) (Experimental)
  Interventions: Biological: Placebo matching with BMS-945429; Biological: BMS-945429
- Induction Cohort: BMS-945429 (Clazakizumab)(400 SC/200 SC mg) (Experimental)
  Interventions: Biological: Placebo matching with BMS-945429; Biological: BMS-945429
- Maintenance Cohort: Placebo matching with BMS-945429 (Clazakizumab) (Experimental)
  Interventions: Biological: Placebo matching with BMS-945429
- Maintenance Cohort: BMS-945429 (Clazakizumab)(100 SC mg) (Experimental)
  Interventions: Biological: BMS-945429
- Maintenance Cohort: BMS-945429 (Clazakizumab)(200 SC mg) (Experimental)
  Interventions: Biological: BMS-945429
- Open Label Cohort: BMS-945429 (Clazakizumab)(200 SC mg) (Experimental)
  Interventions: Biological: BMS-945429

INTERVENTIONS:
Biological: Placebo matching with BMS-945429 — Injection, Intravenous (IV), 0 mg, Day One Only, One Day
  Arms: Induction Cohort: BMS-945429 (Clazakizumab)(400 SC/200 SC mg); Induction Cohort: Placebo matching with BMS-945429 (Clazakizumab)
Biological: Placebo matching with BMS-945429 — Injection, Subcutaneous (SC), 0 mg, Every 4 weeks, 8 weeks
  Arms: Induction Cohort: Placebo matching with BMS-945429 (Clazakizumab)
Biological: Placebo matching with BMS-945429 — Injection, Subcutaneous (SC), 0 mg, Week 4 Only, One Day
  Arms: Induction Cohort: BMS-945429 (Clazakizumab)(150 IV/100 SC mg); Induction Cohort: BMS-945429 (Clazakizumab)(300 IV/100 SC mg); Induction Cohort: BMS-945429 (Clazakizumab)(600 IV/200 SC mg)
Biological: Placebo matching with BMS-945429 — Injection, Subcutaneous (SC), 0 mg, Every 4 weeks, Up to 48 weeks
  Arms: Maintenance Cohort: Placebo matching with BMS-945429 (Clazakizumab)
Biological: BMS-945429 — Injection, Intravenous (IV), 600 mg, Day One Only, One Day
  Other Names: Clazakizumab
  Arms: Induction Cohort: BMS-945429 (Clazakizumab)(600 IV/200 SC mg)
Biological: BMS-945429 — Injection, Subcutaneous (SC), 200 mg, Week 8 only, One Day
  Other Names: Clazakizumab
  Arms: Induction Cohort: BMS-945429 (Clazakizumab)(400 SC/200 SC mg); Induction Cohort: BMS-945429 (Clazakizumab)(600 IV/200 SC mg)
Biological: BMS-945429 — Injection, Intravenous (IV), 300 mg, Day One Only, One Day
  Other Names: Clazakizumab
  Arms: Induction Cohort: BMS-945429 (Clazakizumab)(300 IV/100 SC mg)
Biological: BMS-945429 — Injection, Subcutaneous (SC), 100 mg, Week 8 Only, One Day
  Other Names: Clazakizumab
  Arms: Induction Cohort: BMS-945429 (Clazakizumab)(150 IV/100 SC mg); Induction Cohort: BMS-945429 (Clazakizumab)(300 IV/100 SC mg)
Biological: BMS-945429 — Injection, Subcutaneous (SC), 400 mg, Day One and Week 4, 4 weeks
  Other Names: Clazakizumab
  Arms: Induction Cohort: BMS-945429 (Clazakizumab)(400 SC/200 SC mg)
Biological: BMS-945429 — Injection, Intravenous (IV), 150 mg, Day One Only, One Day
  Other Names: Clazakizumab
  Arms: Induction Cohort: BMS-945429 (Clazakizumab)(150 IV/100 SC mg)
Biological: BMS-945429 — Injection, Subcutaneous (SC), 100 mg, Every 4 weeks, Up to 48 weeks
  Other Names: Clazakizumab
  Arms: Maintenance Cohort: BMS-945429 (Clazakizumab)(100 SC mg)
Biological: BMS-945429 — Injection, Subcutaneous (SC), 200 mg, Every 4 weeks, Up to 48 weeks
  Other Names: Clazakizumab
  Arms: Maintenance Cohort: BMS-945429 (Clazakizumab)(200 SC mg)
Biological: BMS-945429 — Injection, Subcutaneous (SC), 200 mg, Every 4 weeks, Up to 96 weeks, depending on when subject enters this period
  Other Names: Clazakizumab
  Arms: Open Label Cohort: BMS-945429 (Clazakizumab)(200 SC mg)

SUMMARY:
The purpose of this study is to characterize the safety, efficacy and dose response of BMS-945429 in subjects with moderate to severe Crohn's disease and who have had an insufficient response to conventional therapy or have failed Anti-Tumor Necrosis Factor (anti-TNF) therapy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Crohn's Disease diagnosis via radiology, endoscopy or histology within prior 12 months. Diagnosed for at least 3 months
* Active Disease with Crohn's Disease Activity Index (CDAI) ≥ 220 and ≤ 450
* Failed conventional therapy or steroid dependent

Exclusion Criteria:

* Diagnosed/clinical findings of Ulcerative Colitis (UC), indeterminate colitis, non colonic/ileal disease
* Stricture/stenosis, Stoma, proctocolectomy, subtotal colectomy, ileorectal anastomosis
* History of diverticulitis, or evidence of Gastrointestinal (GI) perforations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (53):
- United States (8):
  - University Of California, San Diego, La Jolla, California
  - Precision Research Institute, Llc, San Diego, California
  - South Denver Gastroenterology, Pc, Lone Tree, Colorado
  - University Of Florida, Gainesville, Florida
  - University Of Louisville, Louisville, Kentucky
  - Premier Medical Group Of The Hudson Valley, Pc, Poughkeepsie, New York
  - Options Health Research, Llc, Tulsa, Oklahoma
  - Gastro One, Germantown, Tennessee
- Local Institution, Vienna, Austria
- Canada (3):
  - Local Institution, Calgary, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Saskatoon, Saskatchewan
- Local Institution, Hradec Králové, Czechia
- France (5):
  - Local Institution, Clermont-Ferrand
  - Local Institution, Lille
  - Local Institution, Nice
  - Local Institution, Pessac
  - Local Institution, Saint-Priest-en-Jarez
- Germany (6):
  - Local Institution, Düsseldorf
  - Local Institution, Frankfurt A. M
  - Local Institution, Herne
  - Local Institution, Kiel
  - Local Institution, Magdeburg
  - Local Institution, Münster
- Local Institution, Hong Kong, Hong Kong
- Hungary (3):
  - Local Institution, Budapest
  - Local Institution, Debrecen
  - Local Institution, Pécs
- India (5):
  - Local Institution, Hyderabad, Andhra Pradesh
  - Local Institution, Mumbai, Maharashtra
  - Local Institution, Ludhiana
  - Local Institution, Mumbai
  - Local Institution, Pune
- Israel (3):
  - Local Institution, Jerusalem
  - Local Institution, Rehovot
  - Local Institution, Tel Aviv
- Italy (5):
  - Local Institution, Florence
  - Local Institution, Padua
  - Local Institution, Roma
  - Local Institution, San Donato Milanese (mi)
  - Local Institution, San Giovanni Rotondo (fg)
- Mexico (2):
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Monterrey, Nuevo León
- Local Institution, Nijmegen, Netherlands
- Poland (3):
  - Local Institution, Krakow
  - Local Institution, Lodz
  - Local Institution, Wroclaw
- Local Institution, Seoul, South Korea
- Local Institution, Zurich, Switzerland
- Taiwan (2):
  - Local Institution, Kaohsiung City
  - Local Institution, Taipei
- United Kingdom (2):
  - Local Institution, Hull, Kingston Upon Hull, City of
  - Local Institution, Harrow

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Intravenous (IV), Day One Only Subcutaneous (SC), Every 4 weeks for 8 weeks
- Clazakizumab (150 IV/100 SC): IV, 150 mg, Day One Only SC, 100 mg, Week 8 Only, One Day
- Clazakizumab (300 IV/100 SC): IV, 300 mg, Day One Only SC, 100 mg, Week 8 Only, One Day
- Clazakizumab (400 SC/200 SC): SC, 400 mg, Day One and Week 4 SC, 200 mg, Week 8 only, One Day
- Clazakizumab (600 IV/200 SC): IV, 600 mg, Day One Only SC, 200 mg, Week 8 Only, One Day
Period: Overall Study
Arm/Group | Placebo | Clazakizumab (150 IV/100 SC) | Clazakizumab (300 IV/100 SC) | Clazakizumab (400 SC/200 SC) | Clazakizumab (600 IV/200 SC)
Started | 18 | 9 | 9 | 18 | 18
Completed | 11 | 4 | 4 | 6 | 9
Not Completed | 7 | 5 | 5 | 12 | 9
Not completed — Lack of Efficacy | 0 | 0 | 0 | 3 | 2
Not completed — Adverse Event | 1 | 1 | 2 | 2 | 0
Not completed — Discontinued study treatment | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 2 | 1
Not completed — Participant no longer meets study criteria | 0 | 2 | 0 | 0 | 1
Not completed — Administrative reason by sponsor | 4 | 2 | 3 | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Clazakizumab (150 IV/100 SC) | Clazakizumab (300 IV/100 SC) | Clazakizumab (400 SC/200 SC) | Clazakizumab (600 IV/200 SC) | Total
Number analyzed (Participants) | 18 | 9 | 9 | 18 | 18 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 9 | 8 | 18 | 17 | 69
  >=65 years | 1 | 0 | 1 | 0 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (11.70) | 36.3 (14.79) | 36.2 (17.29) | 36.3 (10.96) | 40.9 (11.48) | 38.6 (12.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 5 | 7 | 10 | 9 | 45
  Male | 4 | 4 | 2 | 8 | 9 | 27

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Clinical Remission (CDAI<150) as Measured by the Crohn's Disease Activity Index (CDAI)
Description: CDAI scores range from 0 to 600. A score of less than 150 corresponds to relative disease quiescence (remission); 150 to 219, mildly active disease; 220 to 450, moderately active disease; and greater than 450, severe disease. A decrease in greater than 100 points indicates a clinically significant improvement in disease activity
Time Frame: At 8 weeks during the Induction Period
Population: modified Intent-to-Treat (mITT) defined as all randomized and treated subjects who had a chance to reach Day 57 by the date of study termination
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Clazakizumab (150 IV/100 SC) | Clazakizumab (300 IV/100 SC) | Clazakizumab (400 SC/200 SC) | Clazakizumab (600 IV/200 SC)
Number analyzed (Participants) | 17 | 9 | 8 | 16 | 16
percentage of participants | 17.6 | 33.3 | 0 | 18.8 | 12.5

2. Secondary Outcome: Percent of Participants With Clinical Response (>100 Point Decrease in CDAI) During Induction Period as Measured by CDAI
Description: as for outcome 1
Time Frame: At 8 weeks during the Induction Period
Population: mITT
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Clazakizumab (150 IV/100 SC) | Clazakizumab (300 IV/100 SC) | Clazakizumab (400 SC/200 SC) | Clazakizumab (600 IV/200 SC)
Number analyzed (Participants) | 17 | 9 | 8 | 16 | 16
percentage of participants | 29.4 | 33.3 | 25.0 | 31.3 | 12.5

3. Secondary Outcome: Change From Baseline at Week 8 and 12 of Inflammatory Bowel Disease Questionnaire (IBDQ) Score
Description: IBDQ consists of 32 questions divided into four dimensions: bowel symptoms (10 items), systemic symptoms (5 items), emotional function (12 items) and social function (5 items). Every question has graded responses from 1 (worst situation) to 7 (best situation), and thus the total score is ranging from 32 to 224 with higher scores representing better quality of life.
Time Frame: Week 8 and Week 12
Population: mITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Clazakizumab (150 IV/100 SC) | Clazakizumab (300 IV/100 SC) | Clazakizumab (400 SC/200 SC) | Clazakizumab (600 IV/200 SC)
Number analyzed (Participants) | 16 | 8 | 8 | 15 | 13
score on a scale
  Week 8: number analyzed (Participants) | 14 | 6 | 8 | 15 | 13
  Week 8 | 11.8 (23.01) | -2.0 (28.93) | 1.9 (36.46) | 15.5 (32.01) | 14.8 (33.7)
  Week 12: number analyzed (Participants) | 14 | 6 | 5 | 8 | 9
  Week 12 | 10.0 (33.65) | 21.8 (34.62) | 1.4 (61.06) | 20.1 (36.32) | 18.7 (35.62)

4. Secondary Outcome: Number of Participants During the Induction Period With Anti-clazakizumab Antibodies
Time Frame: Up to Week 12
Population: mITT
Measure: Number; unit: participants
Arm/Group | Placebo | Clazakizumab (150 IV/100 SC) | Clazakizumab (300 IV/100 SC) | Clazakizumab (400 SC/200 SC) | Clazakizumab (600 IV/200 SC)
Number analyzed (Participants) | 17 | 9 | 9 | 17 | 16
participants | 0 | 0 | 0 | 0 | 1

5. Secondary Outcome: Steady-state Trough Concentration (Cmin) of Clazakizumab During the Induction Period
Time Frame: Week 4, Week 8
Population: Due to early termination of the study, only a limited number of PK samples were collected and analyzed.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Clazakizumab (150 IV/100 SC) | Clazakizumab (300 IV/100 SC) | Clazakizumab (400 SC/200 SC) | Clazakizumab (600 IV/200 SC)
Number analyzed (Participants) | 0 | 0 | 18 | 0
ug/mL
  Week 4: number analyzed (Participants) | 0 | 0 | 17 | 0
  Week 4 |  |  | 21.0816 (8.19326) |
  Week 8: number analyzed (Participants) | 0 | 0 | 8 | 0
  Week 8 |  |  | 36.1026 (14.49349) |

6. Secondary Outcome: Observed Maximum Concentration (Cmax) of Clazakizumab During the Induction Period
Time Frame: Week 0 and Week 4
Population: The interpretation of the PK analysis is limited for several reasons. First, the concentration data that was collected only allowed for reporting of Cmin concentrations. Second, the sample size was limited.
Arm/Group | Clazakizumab (150 IV/100 SC) | Clazakizumab (300 IV/100 SC) | Clazakizumab (400 SC/200 SC) | Clazakizumab (600 IV/200 SC)
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Area Under the Plasma Concentration-time Curve in One Dosing Interval [AUC(TAU)] of Clazakizumab During the Induction Period
Time Frame: Week 0, Week 4, Week 8
Population: as for outcome 6
Arm/Group | Clazakizumab (150 IV/100 SC) | Clazakizumab (300 IV/100 SC) | Clazakizumab (400 SC/200 SC) | Clazakizumab (600 IV/200 SC)
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 12 weeks per participant
Arm/Group | Placebo | Clazakizumab (150 IV/100 SC) | Clazakizumab (300 IV/100 SC) | Clazakizumab (400 SC/200 SC) | Clazakizumab (600 IV/200 SC)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/9 | 1/9 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 2/18 | 2/9 | 2/9 | 6/18 | 4/18
Other Adverse Events (participants affected / at risk) | 1/18 | 2/9 | 3/9 | 8/18 | 2/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=18) | Clazakizumab (150 IV/100 SC) (N=9) | Clazakizumab (300 IV/100 SC) (N=9) | Clazakizumab (400 SC/200 SC) (N=18) | Clazakizumab (600 IV/200 SC) (N=18)
Cronh's disease (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 3
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Anorectal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Anal fistula infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pelvic abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=18) | Clazakizumab (150 IV/100 SC) (N=9) | Clazakizumab (300 IV/100 SC) (N=9) | Clazakizumab (400 SC/200 SC) (N=18) | Clazakizumab (600 IV/200 SC) (N=18)
Injection site erythema (General disorders) | 0 | 0 | 0 | 2 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 2 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site induration (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin depigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Insomnia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Monocyte count increased (Investigations) | 0 | 0 | 0 | 1 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 1 | 0
Protein total decreased (Investigations) | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The interpretation of the PK analysis is limited for several reasons. First, the concentration data that was collected only allowed for reporting of Cmin concentrations. Second, the sample size was limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No